CLINICAL TRIAL: NCT05176327
Title: A Pilot Randomized Controlled Study of the Effects of Exoskeleton Training on Neurogenic Bowel Dysfunction in Spinal Cord Injury/ Disease
Brief Title: Exoskeleton Neurogenic Bowel Dysfunction Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW 21-406
Record Dates: First submitted 2021-12-14; First posted 2022-01-04 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2021-12

CONDITIONS: Spinal Cord Injuries; Neurogenic Bowel
Keywords: spinal cord injuries; neurogenic bowel; exoskeleton; rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries; Neurogenic Bowel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intervention (Experimental): Subjects will receive 2 consecutive courses of exoskeleton training with twelve 45-minute sessions, each to be completed in 6 to 8 weeks. The total period of training will be 12 to 16 weeks.
  Interventions: Device: Exoskeleton training with Ekso NR
- Control (Active Comparator): Subjects will receive twelve 45-minute sessions of usual physiotherapy treatment, consisting of maintenance exercise in the first 6 to 8 weeks, and then one course of exoskeleton training with twelve 45-minute sessions in the following 6 to 8 weeks.
  Interventions: Device: Exoskeleton training with Ekso NR

INTERVENTIONS:
Device: Exoskeleton training with Ekso NR — Walking exercise with Ekso NR

SUMMARY:
The purpose of the study is to assess the effects of exoskeleton training on neurogenic bowel disorders in spinal cord injury/ disease.

DETAILED DESCRIPTION:
After being informed about the study and the potential risks, all patients giving written consents will undergo a medical examination to ensure they are eligible and fit to proceed for the study. Subjects will be randomly assigned to intervention group and control group.

Intervention group will receive 2 consecutive courses of exoskeleton training (ET) with twelve 45-minute sessions, each to be completed in 6 to 8 weeks. The total period of training will be 12 to 16 weeks.

Control group will receive twelve 45-minute sessions of usual physiotherapy treatment (PT), consisting of maintenance exercise in the first 6 to 8 weeks, and then one course of ET with twelve 45-minute sessions in the following 6 to 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. SCI/D for a duration ≥ 12 months
2. Neurological level of injury (NLI) C4 to L3 as defined in the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) 2019 revision
3. Bowel opening via anal route or stoma
4. Stable medical condition
5. Stable mental condition
6. No active painful musculoskeletal problems like fracture, infection, pressure injury, contracture or uncontrolled spasticity
7. Age ≥ 18 years old
8. Body height 150 - 188cm

Exclusion Criteria:

1. Unstable cardiovascular or pulmonary conditions
2. Untreated thromboembolic events
3. Untreated psychiatric disorders
4. History of malignancy
5. Any contra-indications for exoskeleton training

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The change in Neurogenic Bowel Dysfunction (NBD) score in International SCI bowel function basic data set (version 2.0) | Week 0 (Pre-training), Week 8, , Week 16, week 24
  Measurement of the change in the NBD score (0-45, 0-6 Very minor, 7-9 Minor, 10-13 Moderate and 14 or more Severe neurogenic bowel dysfunction) calculated in the data set.

SECONDARY OUTCOMES:
The change in defaecation time (DT) | Week 0 (Pre-training), Week 8, , Week 16, week 24
  The change in average time in minutes to complete defaecation in one week
The change in frequency of bowel incontinence episodes | Week 0 (Pre-training), Week 8, , Week 16, week 24
  The change in number of times of bowel incontinence in the week before

CONTACTS AND LOCATIONS:
Overall Officials: Chor-yin Lam, MBBS, Principal Investigator — The University of Hong Kong
Locations (1):
- MacLehose Medical Rehabilitation Centre, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Sharing of the study protocol, SAP and ICF will be done on request by email to the PI
Supporting Information: Study Protocol, SAP, ICF
Time Frame: From 1 Jan 2024, for a period of 3 years
Access Criteria: On request by email to the PI

REFERENCES:
- [Background] Glickman S, Kamm MA. Bowel dysfunction in spinal-cord-injury patients. Lancet. 1996 Jun 15;347(9016):1651-3. doi: 10.1016/s0140-6736(96)91487-7. PMID 8642958
- [Background] Bloemen-Vrencken JH, Post MW, Hendriks JM, De Reus EC, De Witte LP. Health problems of persons with spinal cord injury living in the Netherlands. Disabil Rehabil. 2005 Nov 30;27(22):1381-9. doi: 10.1080/09638280500164685. PMID 16321920
- [Background] Burns AS, St-Germain D, Connolly M, Delparte JJ, Guindon A, Hitzig SL, Craven BC. Phenomenological study of neurogenic bowel from the perspective of individuals living with spinal cord injury. Arch Phys Med Rehabil. 2015 Jan;96(1):49-55. doi: 10.1016/j.apmr.2014.07.417. Epub 2014 Aug 27. PMID 25172370
- [Background] Benevento BT, Sipski ML. Neurogenic bladder, neurogenic bowel, and sexual dysfunction in people with spinal cord injury. Phys Ther. 2002 Jun;82(6):601-12. PMID 12036401
- [Background] Stiens SA, Bergman SB, Goetz LL. Neurogenic bowel dysfunction after spinal cord injury: clinical evaluation and rehabilitative management. Arch Phys Med Rehabil. 1997 Mar;78(3 Suppl):S86-102. doi: 10.1016/s0003-9993(97)90416-0. PMID 9084372
- [Background] Kinnett-Hopkins D, Mummidisetty CK, Ehrlich-Jones L, Crown D, Bond RA, Applebaum MH, Jayaraman A, Furbish C, Forrest G, Field-Fote E, Heinemann AW. Users with spinal cord injury experience of robotic Locomotor exoskeletons: a qualitative study of the benefits, limitations, and recommendations. J Neuroeng Rehabil. 2020 Sep 11;17(1):124. doi: 10.1186/s12984-020-00752-9. PMID 32917287
- [Background] Miller LE, Zimmermann AK, Herbert WG. Clinical effectiveness and safety of powered exoskeleton-assisted walking in patients with spinal cord injury: systematic review with meta-analysis. Med Devices (Auckl). 2016 Mar 22;9:455-66. doi: 10.2147/MDER.S103102. eCollection 2016. PMID 27042146
- [Background] Esquenazi A, Talaty M, Packel A, Saulino M. The ReWalk powered exoskeleton to restore ambulatory function to individuals with thoracic-level motor-complete spinal cord injury. Am J Phys Med Rehabil. 2012 Nov;91(11):911-21. doi: 10.1097/PHM.0b013e318269d9a3. PMID 23085703
- [Background] Zeilig G, Weingarden H, Zwecker M, Dudkiewicz I, Bloch A, Esquenazi A. Safety and tolerance of the ReWalk exoskeleton suit for ambulation by people with complete spinal cord injury: a pilot study. J Spinal Cord Med. 2012 Mar;35(2):96-101. doi: 10.1179/2045772312Y.0000000003. Epub 2012 Feb 7. PMID 22333043
- [Background] ASIA and ISCoS International Standards Committee. The 2019 revision of the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI)-What's new? Spinal Cord. 2019 Oct;57(10):815-817. doi: 10.1038/s41393-019-0350-9. Epub 2019 Sep 17. No abstract available. PMID 31530900
- [Background] American Spinal Injury Association. International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) (Revised 2019). 2019.
- [Background] Faul F, Erdfelder E, Buchner A, Lang AG. Statistical power analyses using G*Power 3.1: tests for correlation and regression analyses. Behav Res Methods. 2009 Nov;41(4):1149-60. doi: 10.3758/BRM.41.4.1149. PMID 19897823
- [Result] Ozisler Z, Koklu K, Ozel S, Unsal-Delialioglu S. Outcomes of bowel program in spinal cord injury patients with neurogenic bowel dysfunction. Neural Regen Res. 2015 Jul;10(7):1153-8. doi: 10.4103/1673-5374.160112. PMID 26330842
- [Result] Baunsgaard CB, Nissen UV, Brust AK, Frotzler A, Ribeill C, Kalke YB, Leon N, Gomez B, Samuelsson K, Antepohl W, Holmstrom U, Marklund N, Glott T, Opheim A, Penalva JB, Murillo N, Nachtegaal J, Faber W, Biering-Sorensen F. Exoskeleton gait training after spinal cord injury: An exploratory study on secondary health conditions. J Rehabil Med. 2018 Sep 28;50(9):806-813. doi: 10.2340/16501977-2372. PMID 30183055
- [Result] Krogh K, Emmanuel A, Perrouin-Verbe B, Korsten MA, Mulcahey MJ, Biering-Sorensen F. International spinal cord injury bowel function basic data set (Version 2.0). Spinal Cord. 2017 Jul;55(7):692-698. doi: 10.1038/sc.2016.189. Epub 2017 Feb 14. PMID 28195229
- [Result] Krogh K, Christensen P, Sabroe S, Laurberg S. Neurogenic bowel dysfunction score. Spinal Cord. 2006 Oct;44(10):625-31. doi: 10.1038/sj.sc.3101887. Epub 2005 Dec 13. PMID 16344850
- [Result] Huang Q, Yu L, Gu R, Zhou Y, Hu C. Effects of robot training on bowel function in patients with spinal cord injury. J Phys Ther Sci. 2015 May;27(5):1377-8. doi: 10.1589/jpts.27.1377. Epub 2015 May 26. PMID 26157223